CLINICAL TRIAL: NCT01859039
Title: Phase 4 Study to Assess the Safety of Nasal Influenza Immunisation in Egg Allergic Children - a Multicentre Observational Study
Brief Title: Safety of Nasal Influenza Immunisation in Egg Allergic Children
Acronym: SNIFFLE
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Imperial College London (Other); Public Health England (Other Government)
Responsible Party: Principal Investigator, Paul Turner, MRC Clinician Scientist in Paediatric Allergy & Immunology, Imperial College London
Other Study IDs: RHM CHI 0659
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Egg Hypersensitivity
Keywords: Egg allergy; Anaphylaxis; Children; Influenza vaccine
MeSH Terms: conditions — Egg Hypersensitivity; Anaphylaxis; Influenza, Human | interventions — FluMist

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Egg allergic children: Administration of Live attenuated influenza vaccine
  Interventions: Biological: Administration of Live attenuated influenza vaccine

INTERVENTIONS:
Biological: Administration of Live attenuated influenza vaccine
  Other Names: Fluenz (EMA approval number EU/1/10/661/002); FluMist

SUMMARY:
Egg allergy is common in early childhood, affecting at least one in 50 preschool children. Influenza ("'flu") vaccines contain egg protein, as the vaccine is cultured in hen's eggs. There is robust data to support the safety of influenza vaccines (containing low or negligible amounts of egg protein) in patients with egg allergy.

A new influenza vaccine, known as LAIV (Live Attenuated Intranasal Vaccine) has recently been approved by a number of licensing boards and is given by a spray into the nose. This new vaccine has been available in the United States for several years and is highly effective and against influenza infection, with an excellent safety profile in children without egg allergy. However, LAIV is also grown in hen's eggs and contains egg protein, and there are NO existing data on the safety of LAIV in egg-allergic children.

The objective of this multicentre study is to assess the safety of intranasal LAIV in egg-allergic children, in order to demonstrate that these children can safely be given the new LAIV within a primary care health environment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 - 17 years old
* Physician-diagnosis of egg allergy

Exclusion Criteria:

* Contraindicated as acutely unwell or current unstable asthma
* Use of asthma reliever medication in last 72 hours
* Recent administration of a medication containing antihistamine within the last 4 days
* Current oral steroid for asthma exacerbation or course completed within last 2 weeks
* Contraindications to ingredient in LAIV (notwithstanding allergy to egg protein)
* Previous allergic reaction to an influenza vaccine
* Children and adolescents who are clinically immunodeficient due to conditions or immunosuppressive therapy such as: acute and chronic leukaemias; lymphoma; symptomatic HIV infection; cellular immune deficiencies; and high-dose corticosteroids.
* Children and adolescents younger than 18 years of age receiving salicylate therapy because of the association of Reye's syndrome with salicylates and wild-type influenza infection.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and young people with egg allergy between 2-17 years old
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Incidence of allergic reaction to nasal influenza vaccination using a Live Attenuated Influenza Vaccine (LAIV) in egg-allergic children | Within 2 hours of vaccine administration

SECONDARY OUTCOMES:
Incidence of delayed symptoms up to 72 hours after nasal influenza vaccination with LAIV in egg-allergic children | 72 hours after vaccine administration

OTHER OUTCOMES:
Incidence of immediate allergic reaction to LAIV in the subgroups described below. | Within 2 hours of vaccine administration
  1. By age group 2-5, 5-11, 12-17 years
  2. children with a previous history of anaphylaxis to egg protein,
  3. children who have reacted previously to airborne traces of egg,
  4. children who have egg allergy but are tolerant of baked egg,
  5. Presence of physician-diagnosed asthma / recurrent wheeze
  6. Presence of active allergic rhinitis to common environmental indoor allergens

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Turner, FRACP PhD, Principal Investigator — Imperial College London; Mich Erlewyn-Lajeunesse, DM FRCPCH, Principal Investigator — University Hospitals Southampton NHS Foundation Trust
Locations (12):
- United Kingdom (12):
  - Sandwell General Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Royal Hospital for Sick Children, Edinburgh
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Children's Hospital, Liverpool
  - Evelina Children's Hospital, London
  - Imperial College Healthcare NHS Trust (St. Mary's Hospital), London
  - London St George's Hospital, London
  - Manchester Royal Children's, Manchester
  - Newcastle Freeman Hospital, Newcastle
  - Oxford, Oxford
  - University Hospitals Southampton NHS Foundation Trust, Southampton

REFERENCES:
- [Result] Turner PJ, Southern J, Andrews NJ, Miller E, Erlewyn-Lajeunesse M; SNIFFLE Study Investigators. Safety of live attenuated influenza vaccine in atopic children with egg allergy. J Allergy Clin Immunol. 2015 Aug;136(2):376-81. doi: 10.1016/j.jaci.2014.12.1925. Epub 2015 Feb 13. PMID 25684279